CLINICAL TRIAL: NCT03565133
Title: The Effect of Quinine on Food Intake: Oral Sham Feeding Versus Intragastric Delivery
Brief Title: Quinine and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: METC183012
Record Dates: First submitted 2018-05-01; First posted 2018-06-21 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will be blinded for the contents of the gastric capsule. Both cannot be blinded for the oral sham feeding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oral quinine, gastric placebo (Experimental): Oral sham feeding of quinine and a gastric capsule containing placebo (cellulose)
  Interventions: Dietary Supplement: Quinine sham feeding quinine; Dietary Supplement: Gastric placebo
- Oral placebo, gastric quinine (Experimental): Oral sham feeding of placebo (tap water) and a gastric capsule containing quinine
  Interventions: Dietary Supplement: Gastric quinine; Dietary Supplement: Oral sham feeding placebo
- Oral quinine, gastric quinine (Experimental): Oral sham feeding of quinine and a gastric capsule containing quinine
  Interventions: Dietary Supplement: Quinine sham feeding quinine; Dietary Supplement: Gastric quinine
- Oral placebo, gastric placebo (Placebo Comparator): Oral sham feeding of placebo (tap water) and a gastric capsule containing placebo (cellulose)
  Interventions: Dietary Supplement: Oral sham feeding placebo; Dietary Supplement: Gastric placebo

INTERVENTIONS:
Dietary Supplement: Quinine sham feeding quinine — Oral sham feeding with quinine
  Arms: Oral quinine, gastric placebo; Oral quinine, gastric quinine
Dietary Supplement: Gastric quinine — A gastric capsule containing quinine
  Arms: Oral placebo, gastric quinine; Oral quinine, gastric quinine
Dietary Supplement: Oral sham feeding placebo — Oral sham feeding with placebo (tap water)
  Arms: Oral placebo, gastric placebo; Oral placebo, gastric quinine
Dietary Supplement: Gastric placebo — A gastric capsule containing placebo (cellulose)
  Arms: Oral placebo, gastric placebo; Oral quinine, gastric placebo

SUMMARY:
Rationale: The appearance of tastants in the small intestine following food ingestion results in the onset of digestion and absorption but can also result in the activation of a negative feedback mechanism from different parts of the intestine to the stomach, the small intestine and to the central nervous system. These processes inhibit food processing, appetite sensations and food intake, and furthermore they increase feelings of satiety and satiation. In this study, we aim to investigate the effects of oral sham feeding and intragastric delivery of a bitter tastant (quinine) on ad libitum food intake, satiation, gastrointestinal symptoms, and heart rate variability.

Objective: To investigate the effect of oral sham feeding and intragastric delivery of a bitter tastant on food intake.

Secondary Objective(s):

1. To compare the effect of oral sham feeding and intragastric delivery of a bitter tastant on satiation.
2. To assess the effect of oral sham feeding and intragastric delivery of a bitter tastant on gastrointestinal symptoms/complaints.
3. To assess the effect of oral sham feeding and intragastric delivery of a bitter tastant on heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* Based on medical history and previous examination, no gastrointestinal complaints and/or gastrointestinal disorders can be defined.
* Age ≥18 and ≤65 years. This study will include healthy adult subjects (male and female).
* BMI ≥18 and ≤25 kg/m2
* Body weight stable over at least the last 6 months (≤ 5% weight change allowed)

Exclusion Criteria:

* History of severe cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/psychiatric diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol. The severity of the disease (major interference with the execution of the experiment or potential influence on the study outcomes) will be decided by the principal investigator.
* Use of medication that can influence study end-points (to be discussed by medical doctor and principal investigator), including vitamin supplementation, within 14 days prior to testing
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study
* Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy and hysterectomy allowed, and other surgery upon judgement of medical doctor and principle investigator)
* Dieting (medically prescribed, vegetarian, diabetic, macrobiological, biological dynamic)
* Unwillingness to eat lasagna Bolognese meal
* Pregnancy, lactation
* Excessive alcohol consumption (>20 alcoholic consumptions per week)
* Smoking
* Non-tasters of bitter

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Ad libitum food intake | on each test day at T= 50, 50 minutes after ingestion of the capsule and sham-feeding
  Difference in ad libitum meal intake (as measured during ad libitum pasta meal)

SECONDARY OUTCOMES:
Satiation/satiety | At T= -20 mins, T= -10 mins, T=0 mins, T= 10 mins, T= 20 mins, T= 30 mins, T= 40 mins, T=50 and T= end, where T= 0 is ingestion of capsule and sham-feeding and T= end is whenever the participant finishes the test meal given at T= 50 mins.
  Difference in satiation/satiety (as measured by VAS 0-100mm). VAS scores for satiety feelings (e.g., satiety, fullness, hunger, prospective feeding, desire to eat, desire to snack) will be measured using Visual Analogue Scales (VAS, 0 to 100 mm) anchored at the low end with the most negative or lowest intensity feelings (e.g., extremely unpleasant, not at all), and with opposing terms at the high end (e.g., extremely pleasant, very high, extreme). Volunteers will be asked to indicate on a line which place on the scale best reflects their feeling at that moment. The scoring forms will be collected immediately so that they cannot be used as a reference for later scorings.
GI-symptoms | At T= -20 mins, T= -10 mins, T=0 mins, T= 10 mins, T= 20 mins, T= 30 mins, T= 40 mins, T=50 and T= end, where T= 0 is ingestion of capsule and sham-feeding and T= end is whenever the participant finishes the test meal given at T= 50 mins.
  Difference in gastro-intestinal symptoms (as measured by VAS 0-100mm). VAS scores for gastrointestinal symptoms (burning, bloating, belching, cramps, colics, warm sensation, sensation of abdominal fullness, nausea, pain and relaxation/tensness) will be measured using Visual Analogue Scales (VAS, 0 to 100 mm) anchored at the low end with the most negative or lowest intensity feelings (e.g., extremely unpleasant, not at all), and with opposing terms at the high end (e.g., extremely pleasant, very high, extreme). Volunteers will be asked to indicate on a line which place on the scale best reflects their feeling at that moment. The scoring forms will be collected immediately so that they cannot be used as a reference for later scorings.
Heart rate variability | At T= -150 mins, T= -15 mins, T= 5 mins, and T= 35 mins, where T= -150 is 150 minutes before ingestion of standardized breakfast meal, T= 0 mins is ingestion of capsule and sham-feeding.
  Difference in heartrate variability

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Venlo, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No